CLINICAL TRIAL: NCT00823108
Title: Rapid Administration of Insulin in Sepsis: A Pilot Study
Brief Title: Rapid Administration of Insulin in Sepsis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 12-08-23B
Record Dates: First submitted 2009-01-14; First posted 2009-01-15 (Estimated); Last update posted 2022-04-25 (Actual); Status verified 2011-05

CONDITIONS: Septic Shock
Keywords: GIK, septic shock, sepsis
MeSH Terms: conditions — Shock, Septic; Sepsis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Glucose-insulin-potassium
  Interventions: Drug: GIK
- 2 (No Intervention): Control

INTERVENTIONS:
Drug: GIK — 12 hour infusion of GIK solution
  Arms: 1

SUMMARY:
The purpose of this study is to determine if a glucose-insulin-potassium (GIK) solution can be safely administered to patients with septic shock. GIK has been used in thousands of critically ill patients in research studies with very few safety concerns. However, there is a lack of data in regards to patients with septic shock. There are many reasons to believe that GIK would be beneficial in sepsis, including improving heart function and decreasing inflammation. This study will administer intravenous GIK for 12 hours continuously and monitor 10 subjects for 24 hours. A control arm will be used and 10 patients will receive the same monitoring but will not receive GIK.

ELIGIBILITY:
Inclusion Criteria:

1. Suspected or confirmed infection;
2. Any two of four criteria of systemic inflammatory response:

   * Temperature > 100.4° or < 96.8° F
   * Heart rate > 90 beats/minute
   * Respiratory rate > 20 breaths/min. or PaCO2 < 32 mm Hg
   * WBC >12,000 or < 4000 cells/µL or > 10% bands
3. Initiation of quantitative resuscitation protocol in the ED;
4. Requirement of high dose vasopressors (defined as a cumulative vasopressor index = 4) to treat shock

Exclusion Criteria:

1. Age <18 years;
2. Pregnancy;
3. Any primary diagnosis other than sepsis;
4. Established Do Not Resuscitate status or advanced directives restricting aggressive care or treating physician deems aggressive care unsuitable;
5. Known hyperkalemia (serum potassium >5.5);
6. Dialysis-dependent renal failure;
7. Anticipated requirement for immediate surgery (within 24 hours);
8. Active participation in another interventional study;
9. Transferred from another hospital setting with sepsis therapy initiated;
10. Inability to obtain informed consent;
11. Cardiopulmonary resuscitation (chest compression or defibrillation) prior to enrollment;
12. Active malignancy currently under treatment (chemo- or radiation therapy);
13. Known systemic allergy to insulin;
14. History of periodic paralysis associated with carbohydrate loading;
15. Receiving continuous intravenous inotropic support (including dobutamine, milrinone, amrinone, and levosimendan).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2009-03; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Absolute safety endpoint (explicit definitions) | During infusion
Change in SOFA score, microcirculatory flow | During infusion

CONTACTS AND LOCATIONS:
Overall Officials: Alan E Jones, MD, Study Director — Carolinas Medical Center
Locations (1):
- Carolinas Medical Center, Charlotte, North Carolina, United States